CLINICAL TRIAL: NCT02676843
Title: Tau PET Imaging With 18F-AV-1451 in Subjects With MAPT Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Edward D Huey, MD, Assistant Professor of Psychiatry and Neurology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAP4551; R01NS076837 (NIH)
Record Dates: First submitted 2016-01-15; First posted 2016-02-08 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Frontotemporal Lobar Degeneration (FTLD); Frontotemporal Dementia (FTD); Tauopathies
Keywords: FTLD; FTD
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Frontotemporal Dementia; Tauopathies | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-AV-1451 (Experimental): Subjects who are microtubule associated protein tau (MAPT) family carriers and non-carriers will receive 18F-AV-1451 by injection, and undergo a Positron Emission Tomography (PET) scan, which will then be qualitatively analyzed to examine tau deposition in the brain.
  Interventions: Drug: 18F-AV-1451

INTERVENTIONS:
Drug: 18F-AV-1451 — A single injection of up to 10 millicuries of 18F-AV-1451 will be administered to subjects, followed by a 20-minute PET scan.
  Other Names: [18F]AV-1451

SUMMARY:
The study will investigate the ability of a new PET tracer, 18F-AV-1451, to detect depositions of a protein, called tau, in the brains of people with a mutation in the tau gene that causes deposition of the protein, and in people without the mutation. Up to three 18F-AV-1451 scans will be performed (one per year) on control subjects without MAPT mutations, presymptomatic mutation carriers, and symptomatic mutation carriers.

DETAILED DESCRIPTION:
Approximately 40% of cases of Frontotemporal lobar Degeneration (FTLD) are also associated with abnormal deposition of tau protein. The purpose of this study is to image MAPT mutation carriers and their non-carrier relatives in order to study the use of this tracer as a biomarker in Frontotemporal Lobar Degeneration with tau deposition (FTLD-tau).

ELIGIBILITY:
Inclusion Criteria:

* Members of families with established MAPT mutations, who either have the capacity to consent to participate in the protocol, or else have designated a surrogate/proxy to consent to participate in this study

Exclusion Criteria:

* Unwillingness to participate
* Usage of medication which significantly prolongs QT interval
* Pregnancy or plans for pregnancy within 90 days after participating in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Huey, MD, Principal Investigator — Columbia University
Locations (1):
- Morton A. Kreitchman PET Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical characteristics subjects such as age, mutation and rating scale/score of mental state in the manuscript.
Time Frame: Availability of the manuscript through journal editors
Access Criteria: Availability of the manuscript through journal editors

RESULTS

PARTICIPANT FLOW:
Groups:
- 18F-AV-1451: Subjects will receive 18F-AV-1451 by injection, and undergo a Positron Emission Tomography (PET) scan, which will then be qualitatively analyzed to examine tau deposition in the brain.
  18F-AV-1451: A single injection of up to 10 millicuries of 18F-AV-1451 will be administered to subjects, followed by a 20-minute PET scan.
Period: Overall Study
Arm/Group | 18F-AV-1451
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18F-AV-1451
Number analyzed (Participants) | 7
Age, Customized [Count of Participants; unit: Participants]
  18-21 years | 0
  22-29 years | 1
  30-39 years | 1
  40-49 years | 0
  50-59 years | 4
  60-69 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: SUVR of 18F-AV-1451
Description: Regional tau deposition will be measured as standardized uptake value ratio (SUVR) of 18F-AV-1451. SUVR (80-100 min post-injection) for 18F-AV-1451 will be calculated two ways: 1) using cerebellar crus as a reference region, and 2) using the Parametric Estimation of Reference Signal Intensity (PERSI) method to create individual white matter reference regions. Binding in the inferior temporal lobe/cortex was used as the primary outcome.
Time Frame: Baseline, 12-month follow up
Population: 5 out of 7 subjects had data collected and analyzed (evaluable repeat imaging after 12 months).
Measure: Median (Full Range); unit: standardized uptake value ratio (SUVR)
Groups:
- 18F-AV-1451 - Non-carriers: Subjects who are microtubule associated protein tau (MAPT) family non-carriers will receive 18F-AV-1451 by injection, and undergo a Positron Emission Tomography (PET) scan, which will then be qualitatively analyzed to examine tau deposition in the brain.
  18F-AV-1451: A single injection of up to 10 millicuries of 18F-AV-1451 will be administered to subjects, followed by a 20-minute PET scan.
- 18F-AV-1451 - Carriers: Subjects who are MAPT family carriers will receive 18F-AV-1451 by injection, and undergo a Positron Emission Tomography (PET) scan, which will then be qualitatively analyzed to examine tau deposition in the brain.
  18F-AV-1451: A single injection of up to 10 millicuries of 18F-AV-1451 will be administered to subjects, followed by a 20-minute PET scan.
Arm/Group | 18F-AV-1451 - Non-carriers | 18F-AV-1451 - Carriers
Number analyzed (Participants) | 2 | 3
standardized uptake value ratio (SUVR)
  Inferior temporal cortex (Cerebellar crus) | 1.07 [0.99 to 1.14] | 1.26 [1.21 to 1.26]
  Inferior temporal cortex (PERSI) | 1.03 [1.01 to 1.05] | 1.34 [1.26 to 1.36]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | 18F-AV-1451
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-AV-1451 (N=7)
Insomnia (General disorders) | 2 (5)
Headache (General disorders) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT02676843/Prot_SAP_000.pdf